CLINICAL TRIAL: NCT05610046
Title: The Impact of Passive Heat Treatment on Glycaemic Response During an Oral Glucose Tolerance Test in Diabetic Patients
Acronym: Sauna-OGTT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: METC 22-057
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Crossover, randomized, controlled trial
Who Masked: Outcomes Assessor
Masking Description: In this trial, neither the participants, nor the researchers who perform the trial days will be blinded to the intervention allocation. However, the researchers performing the blood analysis are blinded to the treatment allocation and are not involved in the research study during the trial days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-heated sauna session (Sham Comparator): The test days will consist of sitting in an infrared sauna cabin (HM-LSE-3 Professional edition, Health Mate, Belgium). Participants will sit in an infrared sauna at 21° Celsius for a total of 40 minutes.
  Interventions: Device: Sham sauna
- Heated sauna session (Experimental): The test days will consist of sitting in an infrared sauna cabin (HM-LSE-3 Professional edition, Health Mate, Belgium). Participants will sit in an infrared sauna at 60° Celsius (humidity not controlled in an infrared sauna) for a total of 40 minutes.
  Interventions: Device: Infrared sauna heating

INTERVENTIONS:
Device: Infrared sauna heating — Participants will sit in an infrared sauna at 60° Celsius (humidity not controlled in an infrared sauna) for a total of 40 minutes.
  Arms: Heated sauna session
Device: Sham sauna — Participants will sit in an inactive infrared sauna at room temperature (21° Celsius) for a total of 40 minutes.
  Arms: Non-heated sauna session

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a metabolic disease with a rapidly increasing incidence world-wide. The disease is characterizedby a decreased glucose tolerance as a result of insulin resistance, resulting in poor blood glycaemic control. Blood glucose loweringmedications are widely available, but their effect stagnates as T2DM progresses. New treatment regimens are required to combatthe disease. Although therapies such as physical exercise have been shown to induce beneficial effects on glycaemic control inT2DM patients, not all patients are able to perform exercise. Passive heating treatment (PHT) might be an alternative strategy toreduce insulin resistance, as it has been postulated to have comparable effects on the cardiovascular system as exercise. PHT hasbeen linked to numerous health benefits, including improved cardiovascular- and pulmonary function, pain alleviation and metabolichealth. In addition, long term use of PHT shows promising effects on glycaemic control in T2DM patients. However, the acute effectsof PHT on glucoregulation are yet to be determined. Therefore, in this study we will assess the acute impact of passive heat treatment on the post-prandial glycaemic response during an OGTT in T2DM patients

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥50 years old
* Body mass index 18.5 - 35 kg/m2
* DM type 2
* Using oral blood glucose lowering medication
* Able to give informed consent

Exclusion Criteria:

* Insulin dependence
* Changes in diabetes medication in the past 3 months
* Allergy for one of the food items used
* >5% weight change in the previous 6 months
* Participating in a structured (progressive) exercise program, or in the past 3 months.
* Frequent (once per week or more) user of infrared (or traditional) sauna in the past 3 months
* Inability to tolerate sauna/high temperatures
* Smoking
* Diagnosed with cardiovascular disease (e.g. unstable angina pectoris or recent myocardial infarction), kidney failure (eGFR < 60 ml/min/1.73m2), rheumatoid arthritis
* Diagnosed musculoskeletal, GI tract, metabolic (except diabetes) or pulmonary (e.g. COPD) disorders that are expected to influence study outcomes
* Having a pacemaker, defibrillator, or any other type of metal implant

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycaemic response (Matsuda index) | 120 minutes
  OGTT

SECONDARY OUTCOMES:
HOMA-IR | Baseline
  fasting glucose and insulin values
Plasma volume/hematocrit | Throughout test day (3h)
Gutt insulin sensitivity index | 120 minutes
  from OGTT values

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, Prof. Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre +, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided